CLINICAL TRIAL: NCT00290225
Title: Controlled Trial of Yoga Breath Based Group Intervention and Client-Centered Exposure Treatment for Relief of Traumatic Stress and Depression in Tsunami Victims
Brief Title: Yoga Breath Program and Client-Centered Exposure for Relief of PTSD in Tsunami Victims
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Victim Services Center, Miami (Other)
Collaborators: National Institute of Mental Health and Neuro Sciences, India (Other); The Art of Living Foundation (Other); India: International Association for Human Values (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VSCIAHVNIMHANS
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: Posttraumatic stress disorder; depression; disaster mental health; yoga; Breathwork; exposure treatments
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Breath Water Sound Course and Traumatic Incident Reduction

SUMMARY:
Study hypothesis: that a standardized course of Eastern practices (Breath Water Sound Course -BWS) will significantly relieve PTSD and depression in tsunami victims. Further, that a client-centered exposure treatment (Traumatic Incident Reduction- TIR) would provide additional, significant relief of PTSD and depression in tsunami victims.

180 tsunami victims in Southern India will be divided into three groups: those that only receive BWS course, those that receive the BWS course and TIR and a wait-list control. They will be pretested with the PCL-17 (PTSD scale), the Beck Depression Inventory and the General Health Questionaire. These scales will also be administered post-service as well as five weeks post pre-testing and at three and six month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Tsunami witness, tsunami victim, and/or lost loved one or property.
2. Ages 18-70
3. Willing to participate for the entire length of this research study.

Exclusion Criteria:

1. Drug addiction, notwithstanding alcohol or tobacco.
2. Schizophrenia or other severe pre-existing mental illness
3. Severe physical disability or illness that would prevent study completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
That the BWS course and TIR will provide significant reduction in scores on the PCL-C, a standardized measure of PTSD symptoms. | improvement in PCL-C scores will occur in one week and persist for the duration of the study: 6 months
That the BWS course and TIR will provide significant relief from clinical depression as measured on BDI. | Improvement in scores on BDI will occur in one week and persist for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vedamurthy Achar, Ph.D., Principal Investigator — National Institute of Mental Health and Neurosciences, India; Teresa Descilo, MSW, Principal Investigator — Victim Services Center, Miami; R. Damodoran, MA, Study Director — International Association for Human Values

REFERENCES:
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya Yogic breathing in the treatment of stress, anxiety, and depression. Part II--clinical applications and guidelines. J Altern Complement Med. 2005 Aug;11(4):711-7. doi: 10.1089/acm.2005.11.711. PMID 16131297
- [Background] Brown RP, Gerbarg PL. Sudarshan Kriya yogic breathing in the treatment of stress, anxiety, and depression: part I-neurophysiologic model. J Altern Complement Med. 2005 Feb;11(1):189-201. doi: 10.1089/acm.2005.11.189. PMID 15750381
- See also: International Association for Human Values — http://www.iahv.org
- See also: Related research to the BWS intervention — http://www.aolresearch.org